CLINICAL TRIAL: NCT02855320
Title: Efficiency of a Nurse-led Self-management Education Intervention in Promoting Safety Knowledge and Skills of Patients With Arthritis Treated Par Biologics
Acronym: BIOSAFE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: K151201
Record Dates: First submitted 2016-07-01; First posted 2016-08-04 (Estimated); Last update posted 2019-01-28 (Actual); Status verified 2018-12

CONDITIONS: Rheumatoid Arthritis (RA); Spondyloarthritis (SpA)
Keywords: Biologics safety; Rheumatoid arthritis; Spondyloarthritis; patient education; self-management
MeSH Terms: conditions — Arthritis, Rheumatoid; Spondylarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PE (patient education) (Experimental): Nurse-led self-management education intervention : The intervention group will benefit from the nurse intervention in addition to usual care : follow up by their rheumatologist in hospital or private care according to usual management of biologics treatment.
  Interventions: Other: Nurse-led self-management education intervention
- Standard (No Intervention): The control group will be followed up by their rheumatologist in hospital or private care according to usual management of biologics treatment.

INTERVENTIONS:
Other: Nurse-led self-management education intervention — A nurse education consultation at M 0 and M3 in addition to the usual care by the rheumatologist. The nurse will assess the patients' health beliefs and educational needs, focusing on safety skills, self-injections and motivation. The control group will have usual care by the rheumatologist.
  Other Names: Nurse-led patient education; Nurse-led patient safety education
  Arms: PE (patient education)

SUMMARY:
Background : Inflammatory arthritis (rheumatoid arthritis (RA) or spondyloarthritis (SpA) are painful chronic diseases which impair quality of life and work capacity. Biologics are very effective and widely used therapies. However, they are known to entail risks, particularly of infections. The risk of severe infections is of 5%/patient-year with a maximum during the first six month after the initiation of the first biologic therapy.

Patient education (PE) is recommended for the management of chronic diseases. In the case of biologics, PE aims to help patients to learn specific skills particularly on safety issues, e.g stopping the biologic treatment in case of fever or surgery. Safety skills are assessed by the validated BIOSECURE questionnaire. PE seems efficient for safety skills in a few non-randomized studies. In 2010 a national cross sectional survey on 677 patients showed that the risk of incorrect answers in the BIOSECURE questionnaire was 4 times lower among patients who had benefited from an education by a nurse or other kind of educational process (OR =3,8 IC95% :[1,68-8,8].

Aims and Hypothesis: this trial aims to investigate the effects of a nurse-led self-management education face to face intervention on safety skills of patients with arthritis treated par sub cutaneous biologics. Our hypothesis is that the intervention group will report better skills at the 6 months follow up compared to usual care i.e information by the rheumatologist in current consultation.

Methods : multicentric randomized controlled open trial with blinded assessment of the primary outcome. The intervention group will have a nurse education consultation at M 0 and M3 in addition to the usual care by the rheumatologist. The nurse will assess the patients' health beliefs and educational needs, focusing on safety skills, self-injections and motivation. The control group will have usual care by the rheumatologist.

DETAILED DESCRIPTION:
Background Inflammatory arthritis (rheumatoid arthritis (RA) or spondyloarthritis (SpA) are painful chronic diseases which impair quality of life and work capacity. Biologics are very effective and widely used therapies. However, they are known to entail risks, particularly of infections, such as pulmonary infections, tuberculosis, and a few cases of opportunist infections.. The risk of severe infections is of 5%/patient-year with a maximum during the first six month after the initiation of the first biologic therapy.

Patient education (PE) is recommended for the management of chronic diseases. In the case of biologics, PE aims to help patients to learn specific skills particularly on safety issues, e.g stopping the biologic treatment in case of fever or surgery. Safety skills are assessed by the validated BIOSECURE questionnaire, a 54 item questionnaire assessing patients competences to deal with fever, infections, vaccination, and other daily life situations ie travelling, surgery, pregnancy. PE seems efficient for safety skills in a few non-randomized studies. In 2010 a national cross sectional survey on 677 patients showed that the risk of incorrect answers in the BIOSECURE questionnaire was 4 times lower among patients who had benefited from an education by a nurse or other kind of educational process (OR =3,8 IC95% :[1,68-8,8]. Although PE is recommended, a small rate of patients are proposed PE : in the national survey only 30% patients had had a face to face nurse consultation and for 11% patients the nurse consultation was part of a self-management program.

When a biotherapy is initiated, the initiation period is known to be critical for the patients motivation, particularly for patients treated by sub cutaneous biotherapy.

Aims and Hypothesis: this trial aims to investigate, as a primary outcome, the effects of a nurse-led self-management education face to face intervention on safety skills of patients with arthritis treated par sub cutaneous biologics. Our hypothesis is that the intervention group will report better skills at the 6 months follow up compared to usual care i.e information by the rheumatologist in current consultation. As the treatment initiation period is of importance, this trial will also include, as secondary outcomes, disease activity coping, patient's quality of life, self-efficacy. Our hypothesis is that the nurse intervention will increase motivation with positive effects on disease activity, patient's quality of life and coping, as well as self-efficacy.

Methods : multicentric randomized controlled open trial with blinded assessment of the primary outcome.

The pre selection visit will take place during the medical consultation. The rheumatologist will check the eligibility criteria. Eligible patients will receive written information and will be invited to participate in the RCT. The pre selection visit and the selection visit will possibly be done during the same medical consultation. At the selection visit a M0, the patients will sign the non-opposition form, will be assessed for baseline characteristics and complete the questionnaires. The randomization schedule will be prepared by the biostatistician using a computer-generated random numbers. The randomization will take place after the medical consultation and completion of the baseline assessment, in order to preserve the blinding. After randomization, the participants will be either in the intervention group (IG) or the control group (CG). Patients of the intervention group will be referred to the nurse, the same day or within 2 weeks ( maximum 4 weeks) after inclusion.

Intervention group. The intervention group will benefit from the nurse intervention in addition to usual care : follow up by their rheumatologist in hospital or private care according to usual management of biologics treatment.

Nurse intervention At M0, the nurse face to face intervention will include 1/ assessment of the patients' health beliefs and educational needs towards arthritis and treatment through a semi directive questionnaire to enhance communication 2/ Information about biologics 3/ specific education on safety skills and self-injections 4/ Motivational communication on biologics treatment. At M3, the nurse will communicate on the patient's experience and motivation and will reinforce the safety messages.

The MO and M3 intervention will last approximately 1 hour 30. The actual duration of the consultation will be left to the nurse's appreciation depending on the patient's needs and will be collected.

The nurse intervention has been standardized through physical meeting among the centers leading to the development of a dedicated educational booklet including : the components of the educational diagnosis, assessment of the patients of educational needs, safety messages and motivational messages. The elaboration of the booklet is derived from previous work on the BIOSECURE study, recommendations for PE and previous work on educational needs of arthritis patients.

All the nurses have been trained for patient education and self-management (University 1 year curriculum or minimum 40 hours training) and specifically for safety issues of biologics.

Control group. The control group will be followed up by their rheumatologist in hospital or private care according to usual management of biologics treatment.

Baseline characteristics

Baseline assessment will include demographics features, age, gender, education level, disease duration, type of arthritis ( RA versus SpA), disease activity measured by the DAS 28 (Disease Activity index) for the patients with RA and the BASDAI ( Bath ankylosing spondylitis disease activity index) for the patients with SpA, comorbidities, patients previous self-reported knowledge, quality of life (SF12), coping and psychological well-being (VASs from the RAID score, AHI Arthritis helplessness index), Disease activity (DAS, ASDAS, BASDAI), beliefs about medication ( BMQ)

Final assessment

Patients of both groups (IG and CG) will be assessed at M6 for primary and secondary outcomes. The administration of the questionnaires will be done by a member of the multidisciplinary team blinded for the treatment group. An additional nurse consultation will be proposed independently to the trial to the patients especially those whose safety knowledge will be proved to be inadequate at M6 assessment.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years
* Patients with RA ( ACR/EULAR criteria), axial or peripheral Spondyloarthritis (ASAS criteria), patients who are eligible for a Sub cutaneous biologic treatment according to the French recommendations of care
* patients naïve from biologics.
* Patients benefiting from French Social Security insurance.

Exclusion Criteria:

* Patients unable to speak or read French language,
* Patients unable to complete a questionnaire or meet with the trial obligations
* Patients suffering from severe cognitive or psychiatric dysfunction

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2017-01-27 (Actual); Primary Completion 2018-11-26 (Actual); Study Completion 2018-11-26 (Actual)

PRIMARY OUTCOMES:
Safety knowledge and skills towards biologic treatment | 6 months
  score of the BIOSECURE Questionnaire, a 54 item questionnaire including competences to deal with fever, infections, vaccination, and other daily life situations

SECONDARY OUTCOMES:
Quality of life | 6 months
  SF12
Severe infections rate | 6 months
  Severe infections will be defined as infections requiring Intravenous antibiotics or hospitalization.
Coping and psychological well-being (RAID Rheumatoid arthritis Impact of disease score) | 6 months
  VASs coping and psychological well-being from the RAID Rheumatoid arthritis Impact of disease score
Coping and psychological well-being (AHI Arthritis helplessness index) | 6 months
  VASs coping and psychological well-being from AHI Arthritis helplessness index
Disease activity (DAS 28) | 6 months
  DAS 28 (Disease Activity index) for the patients with RA
Disease activity (ASDAS) | 6 months
  ASDAS (Ankylosing spondylarthritis Disease activity score) for the patients with SpA
Disease activity (BASDAI) | 6 months
  BASDAI (Bath Ankylosing spondylarthritis Disease activity Index) for the patients with SpA
Beliefs about biologics | 6 months
  BMQ Beliefs about medicine questionnaire (specific)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine BEAUVAIS, Dr, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Service de Rhumatologie Hôpital Saint Antoine, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Beauvais C, Fayet F, Rousseau A, Sordet C, Pouplin S, Maugars Y, Poilverd RM, Savel C, Segard V, Godon B, L'amour C, Perdriger A, Brin F, Peyrard P, Chalier F, Pallot-Prades B, Tuffet S, Griffoul I, Gossec L. Efficacy of a nurse-led patient education intervention in promoting safety skills of patients with inflammatory arthritis treated with biologics: a multicentre randomised clinical trial. RMD Open. 2022 Mar;8(1):e001828. doi: 10.1136/rmdopen-2021-001828. PMID 35296528